CLINICAL TRIAL: NCT01443923
Title: An Open Label, On-Treatment Trial to Assess the Effect of HIV-1 Coinfection on Therapeutic Responses Using Boceprevir, Peg-Interferon-alfa-2b and Ribavirin in HCV Genotype 1, IFN Treatment-Naive Subjects With or Without HIV-1
Brief Title: Boceprevir Drug Combination for Hepatitis C Treatment in People With and Without HIV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to complete enrollment due to newly approved treatment options.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110253; 11-I-0253
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis; HIV/AIDS
Keywords: Hepatitis; Immunological Response; Virological Response; Resistance Mutations; Viral Kinetics; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis; Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Ribavirin

ARMS (2):
- 1-HCV (Active Comparator): Hepatitis C Mono-infected
  Interventions: Drug: Boceprevir; Drug: Peg-Interferon-alfa 2B; Drug: Ribavirin
- 2 HCV/HIV (Active Comparator): Hepatitis C and HIV co-Infected
  Interventions: Drug: Boceprevir; Drug: Peg-Interferon-alfa 2B; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir
Drug: Peg-Interferon-alfa 2B
Drug: Ribavirin

SUMMARY:
Background:

- Standard treatment for the hepatitis C virus (HCV) is a combination of the drugs peg-IFN and ribavirin. However, this treatment is not very effective in people with a serious type of HCV (HCV genotype 1) and also in people who have human immunodeficiency virus (HIV) coinfection. Researchers want to add a new drug, boceprevir to see if it can improve treatment results in people with both HCV genotype 1 and HIV. Boceprevir used in combination with peg-IFN and ribavirin has been recently approved for the treatment of people with HCV genotype 1 infection only, and is currently being studied in those with HIV and HCV.

Objectives:

- To test boceprevir, peg-IFN, and ribavirin as a treatment for HCV genotype 1 in people with HCV monoinfection compared to those with both HIV and HCV infections.

Eligibility:

* Individuals at least 18 years of age who have HCV genotype 1 infection, and have not received interferon treatment for HCV
* Half of the study participants will also have HIV infection.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests.
* Participants will also have heart and liver function tests, and answer questions about mood and depression.
* Those in the study will receive ribavirin tablets to take twice a day, and peg-IFN to inject under the skin weekly.
* Two weeks after starting treatment, participants will have blood tests to study the treatment.
* Four weeks after starting treatment, participants will start taking boceprevir three times a day.
* Participants will have regular study visits with blood samples and other tests. The length of therapy will depend on the level of virus detected in the blood at several clinic visits. Those who do not respond well to the medicines at 12 weeks will stop treatment. The full length of treatment is 48 weeks.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the United States, an estimated 4.1 million people are infected and HCV is the principal cause of death from liver disease and leading indication for liver transplantation. A combination of ribavirin (RBV) and pegylated interferon (peg-IFN) is the currently recommended therapy for chronic HCV infection. However, this therapy achieves viral clearance in only 19% to 52% of patients infected with HCV genotype 1 and 76% to 80% of patients infected with genotypes 2 and 3. Current therapy is also associated with a high incidence of adverse events and low cure rates in several populations. Novel therapies that do not rely on an interferon backbone will be required to enhance cure rates in various populations. Recent data show that adding an HCV serine protease inhibitor (such as boceprevir [BOC]) to peg-IFN and RBV results in HCV eradication rates of 70% to 80% among HCV-monoinfected subjects. However, whether human immunodeficiency virus (HIV)-infected subjects will have similar rates of response to triple combination therapy is presently not known. Previous data have suggested that HIV-infected patients with chronic HCV infection have much lower eradication rates to peg-IFN and RBV than HCV-monoinfected subjects. This study will explore whether HIV/HCV-coinfected subjects have a lower response rate to a BOC/peg-IFN/RBV regimen than HCV-monoinfected subjects. Participants who have chronic hepatitis C genotype 1 monoinfection (N=50) or coinfection with HIV-1 (N=50), and who are na(SqrRoot) ve to IFN-based HCV treatment, will receive combination therapy with BOC (800 mg three times a day, every 7 to 9 hours, with food), weekly peg-IFN alpha-2b (1.5 mcg/kg/week) and twice daily RBV (weight based) for a maximum of 44 weeks, after a 4-week lead-in of peg-IFN and RBV. BOC received recent FDA approval for treating HCV monoinfection in combination with peg-IFN and RBV, and the approved labeling will be followed in this study. The primary endpoint is comparative efficacy in HCV-monoinfected and HIV/HCV-coinfected subjects. Secondary endpoints include determination of host predictors for therapeutic response, emergence of resistance biomarkers, and early viral kinetics. The findings from this study will aid in the understanding of whether HIV infection affects HCV antiviral and host responses to combination therapy using BOC/peg-IFN alfa-2b/RBV.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for participation on this protocol, a participant must satisfy all of the following conditions:

1. Be greater than or equal to18 years old and have an identifiable primary care provider.
2. Have documented chronic HCV infection by demonstration of a positive test for hepatitis C antibody and HCV RNA of 2,000 IU/mL or greater.
3. Infected with HCV GT-1 virus.
4. If coinfected, have either documentation of HIV-1 infection by licensed enzyme-linked immunosorbent assay (ELISA) confirmed by a Western Blot or history of HIV RNA of 1,000 copies/mL or greater.
5. If coinfected, must meet one of the following prior to enrollment:

   1. If on a stable non-NNRTI or non-PI antiretroviral regimen that HAS NOT changed within the past 6 months, must have an HIV-1 VL of less than 400 copies/mL for at least 3 months; or
   2. If on a current antiretroviral regimen that HAS changed within the past 6 months, have an HIV-1 VL of less than 50 copies/mL for at least 3 months; or
   3. Be a long-term nonprogressor as documented in the medica record.
6. Have histopathologic features consistent with chronic HCV infection at the time of enrollment. A liver biopsy within 3 years (36 calendar months) prior to screening may be used as the baseline biopsy. Participants can opt out of a liver biopsy if they had one more than 3 years prior and have a contraindication, such as receipt of chronic anticoagulation therapy. Participants with decompensated liver disease are excluded from the study.
7. Are na(SqrRoot) ve to prior IFN-based treatment for HCV.
8. Have CD4 cell counts greater than or equal to 100 cells/mm(3).
9. Willing to have genetic testing.
10. Not pregnant or breastfeeding. Serum pregnancy test must be negative at screening for female participants.
11. Agree not to become pregnant if a female of childbearing potential while on the study and for at least 6 months after stopping RBV. Because of the potential teratogenic effects of RBV treatment, subjects and their partners must remain abstinent or use two methods of birth control, which may be selected from the following list (oral contraceptive concentrations are decreased, and may not be effective when used during BOC treatment and, therefore, are not included in this list):

    Surgical sterilization of either partner

    Intrauterine device

    Male or female condoms with or without a spermicide

    Diaphragm, cervical cap, or sponge
12. Male participants who are not documented to be sterile must agree to either abstain from intercourse or consistently use a condom while their female partner (if applicable) agrees to use one of the appropriate medically accepted methods of birth control listed above from the date of screening until 6 months after the last dose of RBV.
13. Be able and willing to either learn to safely inject medication or find another person to inject the medication for him/her.
14. Be willing to allow storage of blood or tissue samples for future research.

Co-enrollment Guidelines:

Participants may be enrolled in other NIH protocols as long as the amount of research blood drawn does not exceed the acceptable NIH guidelines and the protocol does not include other experimental therapies (including expanded access/compassionate use of HIV antiretrovirals).

EXCLUSION CRITERIA:

A participant will be ineligible to participate on this study if any of the following criteria are met:

1. Use of other experimental therapies (including expanded access/compassionate use of HIV antiretrovirals) within 30 days or 5 half-lives (whichever is longer), prior to enrollment.
2. Current use of an efavirenz-based (or other NNRTI) or protease inhibitor HIV antiretroviral regimen.
3. Use of any of the following medications within 6 weeks prior to enrollment.

   Alfuzosin (Uroxatral )

   Alprazolam (Xanax )

   Atorvastatin (Lipitor )

   AZT or zidovudine (Retrovir )

   Carbamazepine (Tegretol )

   Cisapride (Propulsid )

   Colchicine (Colcrys ) - If patient has renal or hepatic impairment.

   DDI or didanosine (Videx )

   d4T or stavudine (Zerit )

   Delaviridine (Rescriptor )

   Digoxin (Lanoxin )

   Dihydroergotamine

   Drosperinone (Yaz )

   Efavirenz (Sustiva )

   Ergonovine (Ergotrate )

   Ergotamine (Cafergot )

   Etravirine (Intelence )

   Ganciclovir (Cytovene )

   Immunosuppressive therapy (including oral steroids)

   ---Use of any use of any immunosuppressive therapy, including systemic steroids (prednisone equivalent of greater than 10 mg/day) for a duration of 6 weeks or more within 6 months prior to enrollment. Use of inhaled/nasal steroids should be avoided.

   Isoniazid or INH (Ingredient in Rifater )

   Ketoconazole (Nizoral )

   Lovastatin (Mevacor )

   Methylergonovine (Methergine )

   Midazolam given orally (Versed )

   Nevirapine (Viramune )

   Phenobarbital (Luminal )

   Phenytoin (Dilantin )

   Pimozide (Orap )

   Pyrazinamide (Ingredient in Rifater )

   Rifabutin (Mycobutin )

   Rifampin/rifampicin

   Rilpivirine (Edurant )

   Sildenafil (Viagra ) - Phosphodiesterase type 5 inhibitors are prohibited when used for pulmonary hypertension

   Simvistatin (Zocor )

   St. Johns s Wort

   Tadalafil (Cialis ) - Phosphodiesterase type 5 inhibitors are prohibited when used for pulmonary hypertension

   Thalidomide (Thalomid )

   Theophylline (Slo-Phylllin )

   Triazolam (Halcion )

   Vardenafil (Levitra ) - Phosphodiesterase type 5 inhibitors are prohibited when used for pulmonary hypertension

   Warfarin (Coumadin )

   Zalcitabine (Hivid )

   There may be other brand names for these products listed above.
4. Has ingested silymarin (milk thistle), s-adenosylmethionine (SAM-e), glycyrrhizin, Sho-saiko-to (SST), or other herbal supplements that may be either liver beneficial or toxic, within 28 days prior to enrollment.
5. Mixed HCV genotypes (e.g., 1 & 2, 1 & 3, 1 & 4) (mixed genotype 1a/1b can be included).
6. Has any other known, or clinically suspected, cause of liver disease, including active hepatitis B.
7. For participants with cirrhosis, a Child Turcotte Pugh score greater than 7, or Child s B or C cirrhosis.
8. Certain abnormal hematological and biochemical parameters, including:

   1. Neutrophil count less than1000 cells/mm3
   2. Hemoglobin less than10g/dL
   3. Platelet count less than or equal to 50,000 cells/mm3
   4. Estimated glomerular filtration rate less than50 mL/min/1.73 m(2), calculated automatically by the NIH lab using the original MDRD (modification of diet in renal disease) study equation
   5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than or equal to10 time ULN
   6. Prothrombin time International Normalized Ratio (PT-INR) less than2 and/or on chronic anticoagulation medications
   7. If total bilirubin is greater than 1.5 mg/dL, then direct bilirubin can be no more than 70% of the total, up to a direct bilirubin of 2.0 mg/dL.
9. Alpha-fetoprotein less than20 ng/mL, unless an ultrasound, computerized tomography scan (CT), or magnetic resonance imaging (MRI) has been performed to rule out hepatoma.
10. Hepatic mass suggestive of hepatocellular carcinoma as detected by ultrasound scan, dual-phase CT, or MRI.
11. History of esophageal or gastric varices.
12. Any neoplastic disease or any nonmetastatic skin, cervical, or anal cancer that has been resected in the past 5 years EXCEPT Kaposi s sarcoma not requiring systemic chemotherapy.
13. Prior organ transplantation other than cornea or hair.
14. Evidence of severe cardiac disease (greater than or equal to Grade 3 congestive cardiac failure, symptomatic coronary artery disease, significant arrhythmias, or uncontrolled hypertension) despite intervention or medical therapy.
15. Evidence of severe chronic pulmonary disease with functional impairment.
16. Severe psychiatric disorder that would interfere with adherence to protocol requirements, and that is not stably treated.
17. Evidence of autoimmune disorders including inflammatory bowel diseases, psoriasis, and optic neuritis.
18. Evidence of an uncontrolled seizure disorder defined as more than 1 episode of generalized seizure within the past year.
19. Chronic pancreatitis based on clinical history.
20. History of severe retinopathy.
21. History of hemophilia.
22. Any hemoglobinopathy (e.g., Thalassemia, sickle cell disease).
23. Active systemic infections other than HCV and HIV-1.
24. Evidence of gastrointestinal malabsorption, chronic nausea, or vomiting.
25. Has any systemic illness that will make it unlikely that the participant will be able to return for the required study visits.
26. Any condition that, in the opinion of the investigator, contraindicates participation in this protocol.

Exclusion of Children:

Because there are insufficient data regarding the safety and efficacy of BOC, PEG, or RBV in the pediatric population, children are excluded from this study.

Exclusion of Women:

Pregnancy: Pregnant women are excluded from this study because the effects of BOC, PEG, and RBV on the developing human fetus are unknown. Preclinical animal data indicate that the use of RBV treatment during pregnancy is potentially teratogenic.

Breastfeeding: Because there is an unknown but potential risk for adverse effects in nursing infants secondary to treatment of the mother with BOC, PEG, or RBV, breastfeeding women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kottilil, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - Unity Health Care, Inc./DC General, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Kim WR. The burden of hepatitis C in the United States. Hepatology. 2002 Nov;36(5 Suppl 1):S30-4. doi: 10.1053/jhep.2002.36791. PMID 12407574
- [Background] Congote LF, Trachewsky D. Qualitative changes in nuclear RNA from rat kidney cortex after aldosterone treatment. Biochem Biophys Res Commun. 1972 Jan 31;46(2):957-63. doi: 10.1016/s0006-291x(72)80234-1. No abstract available. PMID 5057920

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-HCV: Hepatitis C Mono-infected
  Boceprevir
  Peg-Interferon-alfa 2B
  Ribavirin
- 2 HCV/HIV: Hepatitis C and HIV co-Infected
  Boceprevir
  Peg-Interferon-alfa 2B
  Ribavirin
Period: Overall Study
Arm/Group | 1-HCV | 2 HCV/HIV
Started | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-HCV | 2 HCV/HIV | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (3) | 56 (0) | 57.5 (2.64575)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Defined as Sustained Viral Response (SVR) Six Months After the End of Specified Treatment.
Time Frame: 6 months post treatment
Population: Due to the change in the standard of care treatment of HCV, it became difficult to recruit patients to receive IFN based therapy with the prospects of IFN free treatment being available sooner. Study was prematurely terminated and no data was collected/analyzed for the Outcome.
Arm/Group | 1-HCV | 2 HCV/HIV
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Early HCV Viral Load Kinetics Between Mono and Co-infected Subjects
Time Frame: Day 0, Day 7
Population: as for outcome 1
Arm/Group | 1-HCV | 2 HCV/HIV
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Safety and Treatment Outcome Measures Stratified by ESA Use
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | 1-HCV | 2 HCV/HIV
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Subjects Who Are Receiving HAART Who Remain With an HIV RNA & lt; 400 Copies/mL and Those With HIV RNA & gt; 400 Copies/mL at End of Treatment
Time Frame: End of Treatment
Population: as for outcome 1
Arm/Group | 1-HCV | 2 HCV/HIV
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Efficacy (SVR) Rates as Predicted by Viral Response at the End of the 4-week lead-in Therapy With PEG/RBV and Comparison Between HCV Monoinfected and HIV/HCV Coinfected Subjects
Time Frame: 6 months post treatment
Population: as for outcome 1
Arm/Group | 1-HCV | 2 HCV/HIV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1-HCV | 2 HCV/HIV
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-HCV (N=3) | 2 HCV/HIV (N=1)
Abdomina Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) — Seizure: (New Onset)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute Kidney Injury
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-HCV (N=3) | 2 HCV/HIV (N=1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Injection Site Reaction (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) — CommonCold
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (8) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) — Seizures
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes